CLINICAL TRIAL: NCT06783348
Title: Phase II Trial Evaluating the Efficacy of 177Lutetium-PSMA-617 Treatment in Patients With Metastatic Clear Cell Renal Carcinoma Cell With Progressive Disease on First-line or Second-line Systemic Treatment
Brief Title: Radiopharmaceutical Treatment of Advanced Kidney Cancer
Acronym: RENALUT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-2361-GUCG; 2024-517899-38-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Clear Cell Renal Cell Carcinoma
Keywords: renal cancer
MeSH Terms: conditions — Clear-cell metastatic renal cell carcinoma; Kidney Neoplasms | interventions — Pluvicto

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): 177Lu-PSMA-617 will be administered by intravenous infusion or injection at an activity of 7.4 GBq every 6 weeks (±1 week) for up to a total of 6 doses, unless there is disease progression or unacceptable toxicity or until the occurrence of a withdrawal criterion. The first infusion should be administered within 3 weeks from enrolment. Patients in PR or SD after 4 cycles will receive an additional two doses.
  Interventions: Drug: 177Lu-PSMA-617

INTERVENTIONS:
Drug: 177Lu-PSMA-617 — Administeration by intravenous infusion or injection at an activity of 7.4 GBq every 6 weeks (±1 week) for up to a total of 6 doses, unless there is disease progression or unacceptable toxicity or until the occurrence of a withdrawal criterion. The first infusion should be administered within 3 weeks from enrolment. Patients in PR or SD after 4 cycles will receive an additional two doses.

SUMMARY:
Background This study is for adults with advanced kidney cancer that has spread to other parts of the body and has continued to progress despite treatment with immunotherapy and targeted therapy. Unfortunately, treatment options at this stage of the disease are limited. The existing treatments' ability to work against cancer has not been fully looked into.

Rationale The goal of this study is to examine if a new drug treatment called 177Lutetium-PSMA-617, hereafter referred as 177Lu-PSMA-617, which holds the active ingredient 177Lutetium-PSMA and has been used as a standard treatment for advanced prostate cancer since December 2022, can also help treat advanced kidney cancer.

The drug 177Lu-PSMA-617 is being tested as an experimental treatment that targets a specific protein on cancer cells. This protein, known as prostate-specific membrane antigen (PSMA), is present on the surface of kidney cancer cells. Therefore, before the treatment begins, participants will undergo a PET (positron-emission tomography) scan to check if their kidney cancer cells express high levels of PSMA. This scan uses a small amount of radioactive material (in the form of 177Lutetium) to visualize the presence of PSMA on the cancer cells. Only participants who test positive for PSMA can take part in the study. In this approach, PSMA serves two purposes. First, it helps assess whether the cancer expresses this protein and allows 177Lu-PSMA-617 to specifically target and attach to the cancer cells. Second, 177Lu-PSMA-617 delivers a small amount of radiation directly to the tumour, which helps kill cancer cells while minimizing damage to normal cells. This type of treatment is known as a radiopharmaceutical.

Objective The primary aims are to find out if 177Lu-PSMA-617 is useful against kidney cancer and to assess its safety. Throughout the study, participants will undergo several imaging assessments to check their disease and response to treatment.

The study also includes the collection of tissue samples. Together with the information collected from the imaging assessments, this will allow further research into markers that may lead to earlier detection of tumour spread or help identify individuals who may benefit more from treatment with 177Lu-PSMA-617.

Treatment All participants will receive 177Lu-PSMA-617 through an intravenous injection at a standard dose of 7,400 MBq (megabecquerel: a measure of radioactivity). Treatments will be administered approximately every six weeks, for a maximum of six times.

Blood tests are done before and during treatment to check the participant's health and to detect any early side effects from the treatment. Different types of scans are performed before, during, and after 177Lu-PSMA-617 administration to check how well the treatment is working. After treatment ends, follow-up visits will be scheduled every six weeks during the first year. In the second year, your doctor will decide how often you need to come in for visits. These appointments are important for monitoring how the body continues to respond to the treatment. The entire study period will last approximately two years from the time of study entry.

Participants

The study will include approximately 56 participants who will be tested for PSMA expression, to obtain a minimum of 48 participants expressing PSMA entering the study. To qualify, participants must:

* Be diagnosed with advanced kidney cancer previously treated with immunotherapy and targeted therapy.
* Test positive for PSMA on a PET scan.
* Be generally healthy and able to perform daily activities.
* Be at least 18 years of age.

Benefit-risk analysis The drug 177Lu-PSMA-617 has proven to work well in treating advanced prostate cancer and could be a promising new treatment possibility for kidney cancer, although this has not yet been shown. By joining this study, participants will contribute to valuable research to better understand kidney cancer and improve treatment options for future patients. Participating in this study offers a chance to try a new treatment, which might help people with advanced kidney cancer live longer and prevent the disease from getting worse, especially for those who have limited treatment options left after immunotherapy and targeted therapy.

With all new treatments, there are possible risks and side effects associated with them. Side effects of the drug 177Lu-PSMA-617 may include feeling tired, nausea, dry mouth, loss of appetite, and changes in blood cells. While not all side effects are known yet, the study team will carefully follow participants for any side effects during and after treatment. It is important to understand that while the study is being done to provide new information, there are still some questions on the treatment's safety and how well it will work.

DETAILED DESCRIPTION:
RATIONALE After progression on first-line Immune Checkpoint Inhibitor (ICI)-based treatment, sequencing of Vascular Endothelial Growth Factor-Receptor Tyrosine Kinase Inhibitors (VEGFR-TKIs) is standard of care as long as the patient derives clinical benefit. Cabozantinib and axitinib, if not given in first line, are good choices in second line. However, the response rate to VEGFR-TKIs in second line remains low, not exceeding 32-41%. In addition, there is no standard of care treatment after ICI- and VEGFR-TKI-based therapy. Therefore, novel therapeutic strategies must be developed.

Given the high efficacy and low toxicity of 177Lu-PSMA-617 reported in prostate cancer, and the observed Prostate-specific Membrane Antigen (PSMA) expression in ccRCC, we propose to evaluate 177Lu-PSMA-617 radioligand therapy (RLT) in metastatic ccRCC patients who progress after treatment with at least one ICI and one VEGFR-TKI given in sequence or in combination in the metastatic setting.

The trial will evaluate 4 cycles of 177Lu-PSMA-617 with 2 additional cycles in case of partial response (PR) or stable disease (SD).

OBJECTIVES The primary objective is to evaluate the activity of 177Lu-PSMA-617 through Objective Response in metastatic ccRCC patients progressing on or after treatment with one ICI, and one VEGFR-TKI, either in combination or in se¬quence.

The secondary objectives are:

* To assess the safety profile of 177Lu -PSMA-617 in patients with metastatic ccRCC
* To estimate disease control rate (DCR), progression-free survival (PFS) and overall survival (OS) of participants with metastatic ccRCC treated with 177Lu-PSMA-617
* To estimate the time to start subsequent systemic treatment for patients with metastatic ccRCC treated with 177Lu-PSMA-617.

The study is a prospective, multicentric, single arm phase II trial.

Number of patients:

Approximately 56 participants will be screened to achieve 48 enrolled to the study intervention and at least 43 to be evaluable for the primary endpoint.

This trial may be beneficial for patients with metastatic RCC progressing after ICI and VEGFR-TKI, for which efficacious alternative treatment options are lacking, and toxicity remains an issue.

These patients will be closely followed with conventional imaging as well as by PSMA-PET/CT, which has been suggested to be more sensitive than conventional imaging in detection of metastases. These patients will be followed in expert centers specialized in renal- and prostate cancer management by physicians experienced in managing progressive mRCC, as well as adverse events related to 177Lu-PSMA-617 treatment.

ELIGIBILITY:
Inclusion Criteria:

PRE-SCREENING

* Histologically proven ccRCC. Sarcomatoid component is allowed.
* Adult patients ≥18 years old.
* Has progressed on or after ≥1-line prior systemic therapy approved in the metastatic setting. Prior treatment must include an anti-programmed death-1 (receptor) [PD-1]/programmed death-ligand 1 (PD-L1) therapy +/- ipilimumab and a VEGFR-TKI.
* Written pre-screening informed consent according to ICH/GCP and local regulations.

SCREENING

* Patients with at least one PSMA-positive metastatic lesion, and no exclusionary PSMA-negative lesions, with positive lesions defined as those with a maximum standardized uptake value (SUVmax) greater than the mean standardized uptake value (SUVmean) of liver background.
* Measurable disease by RECIST 1.1 criteria.
* Patients with adequate blood tests (Absolute neutrophil count > 1.5 x 109/L, haemoglobin > 9.0 g/dL, platelet count > 100,000/µL, estimated glomerular filtration rate (GFR) ≥ 40 ml/min by CKD-EPI formula, total bilirubin ≤ 1.5 x ULN. Aspartate aminotransferase and alanine aminotransferase ≤ 2.5 x ULN (≤ 5 x ULN in patients with liver metastases).
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Women of childbearing potential (WOCBP) must have a negative serum (or urine) pregnancy test within 72 hours prior to registration. A positive urine pregnancy test result must immediately be confirmed using a serum test. A pregnancy test is to be reported within 7 days prior to the first dose of the study treatment.

Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e., females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrhoeic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antioestrogens, low body weight, ovarian suppression, or other reasons.

* Patients of childbearing / reproductive potential should use adequate birth control measures during the study treatment period and for at least 14 weeks after the last dose of treatment. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Such methods include:

  * Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomized partner
  * Sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
  * Female subjects who are breast feeding should discontinue nursing prior to the first dose of study treatment and until 3 months after the last study treatment.
* Before patient's enrolment, written informed consent must be given according to ICH/GCP, and national/local regulations. This includes consent to comply to recommended radioprotection precautions during study.

Exclusion Criteria:

* Patient with RCC in a single kidney.
* Patients with PSMA-negative lesions (defined as PSMA uptake equal to or lower than that of liver parenchyma) in any lymph node with a short axis of at least 15 mm, in any metastatic solid-organ lesions with a short axis of at least 1.0 cm, or in any metastatic bone lesion with a soft-tissue component of at least 1.0 cm in the short axis. Patients with any PSMA-negative metastatic lesion meeting these criteria are ineligible.
* Other malignancy that is expected to interfere with the treatment or results of this study, such as prostate cancer.
* Patient with active uncontrolled or symptomatic central nervous system (CNS metastases).

Note: patients treated previously with radiotherapy and/or surgery resulting in controlled/asymptomatic CNS disease are allowed.

* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be assessed and discussed with the patient before the enrolment in the in the trial.
* Known contraindication to imaging tracer or any product of contrast media.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2028-01-30 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response | 9 months after Last Patient In
  Objective Response, defined as a Complete Response (CR) or a Partial Response (PR) based on RECIST 1.1 criteria, on conventional imaging.

SECONDARY OUTCOMES:
safety (adverse events) | 42 months after First Patient In
  Safety in all treated patients using Common Terminology Criteria for Adverse Events (CTCAE) V5.0
Disease control rate (DCR) at 6-months | 6 months after treatment initiation
  Disease control according to RECIST 1.1 at 6 months (defined as 24 weeks +/- 1 week) after treatment initiation.
Progression-free survival (PFS) | 42 months after First Patient In
Time to start of next systemic treatment | 42 months after First Patient In
  the overall time in months until the patient began the next systemic treatment
Overall survival (OS) | 42 months after First Patient In

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Seront, MD, Principal Investigator — Cliniques Universitaires de Saint Luc

REFERENCES:
- [Derived] Seront E, Bsilat M, Goffin K, Govaerts AS, Litiere S, Cabrieto J, Dhondt B, Tombal B, Albiges L; EORTC Genito-Urinary Cancer Group. Efficacy of [177Lu]Lu-PSMA-617 in Patients with Metastatic Clear-cell Renal Cell Carcinoma: The Multicentre, Single-arm, Phase 2 RENALUT Trial. Eur Urol Oncol. 2025 Dec;8(6):1592-1597. doi: 10.1016/j.euo.2025.09.003. Epub 2025 Oct 10. PMID 41073165